CLINICAL TRIAL: NCT06512753
Title: The Effectiveness of Hydroxychloroquine Versus Methotrexate in the Treatment of Lichen Planopilaris in Routine Clinical Care: a Patient Preference Trial
Acronym: HEMLET
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, DirkJan Hijnen, MD, PhD, Erasmus Medical Center
Other Study IDs: 11940
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Lichen Planopilaris; Cicatricial Alopecia
Keywords: Lichen planopilaris; Cicatricial alopecia; Hydroxychloroquine; Methotrexate
MeSH Terms: conditions — Lichen Planus; Alopecia | interventions — Hydroxychloroquine; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hydroxychloroquine (HCQ): HCQ is administered orally at a dosage of 400 mg daily.
  Interventions: Drug: Hydroxychloroquine
- Methotrexate (MTX): MTX is given at a dose of 15 mg per week, orally or subcutaneously. Additionally, folate supplementation is administered concurrently as part of standard care, with folate 10 mg/week administered 24 hours after MTX intake.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Hydroxychloroquine — HCQ (15) is administered orally at a dosage of 400 mg daily.
  Groups: Hydroxychloroquine (HCQ)
Drug: Methotrexate — MTX (16) is given at a dose of 15 mg per week, orally or subcutaneously. Additionally, folate supplementation is administered concurrently as part of standard care, with folate 10 mg/week administered 24 hours after MTX intake.
  Groups: Methotrexate (MTX)

SUMMARY:
Rationale Lichen planopilaris (LPP) is a prevalent form of cicatricial alopecia, predominantly affecting women and causing irreversible hair loss. Hydroxychloroquine (HCQ) and methotrexate (MTX) are the most frequently used systemics for treatment of LPP in daily practice. Due to the absence of well-established treatment guidelines, this study aims to evaluate the effectiveness of HCQ and MTX in routine clinical care.

Objective(s) To investigate the effectiveness of HCQ and MTX in the treatment of adults with lichen planopilaris in routine clinical care.

Study type Prospective, patient preference clinical trial with a duration up to 48 weeks in accordance with the routine clinical care guidelines.

Study population This study will include adults (≥18 years) diagnosed with LPP.

Methods Patients will choose between HCQ and MTX treatment as in routine clinical care, receiving follow-up in accordance with standard clinical practices. They will not be randomized. The primary endpoint is the measurement of the Lichen Planopilaris Activity Index (LPPAI) at the 6-months, providing a quantitative assessment of the disease's activity and response to the selected treatment. The Skindex-29 questionnaire will be conducted at each visit, allowing evaluation of the impact on patients' quality of life.

DETAILED DESCRIPTION:
Treatment of LPP remains a challenge due to limited evidence-based guidelines and a lack of randomized controlled trials, leading to the absence of standardized therapeutic protocols and outcome measures. Currently, the treatment goal for LPP primarily focuses on halting disease progression to minimize further hair loss and alleviate associated symptoms. Treatment options for LPP include topical/intralesional corticosteroids, and systemic therapies such as hydroxychloroquine (HCQ), methotrexate (MTX), and other immunosuppressive agents. However, the absence of daily practice studies makes it challenging to establish therapeutic recommendations.

This patient preferred trial aims to fill a crucial knowledge gap in LPP management. Existing evidence lacks comprehensive guidelines for treating LPP effectively, leaving current approaches largely empirical. Aligning with the urgent need for answers highlighted by the 'Nederlandse Vereniging voor Dermatologie en Venereologie Kennisagenda Dermatologie 2019': 'Q9 - Wat is de effectiviteit van systemische behandeling bij patiënten met cicatriciële alopeciëen?' (What is the most effective systemic treatment for cicatricial alopecias) (13) underscores the pressing concern regarding the effectiveness of systemic therapy in cicatricial alopecia. This study seeks to contribute novel insights to the field by comparing the effectiveness of the two most commonly used systemic treatments, HCQ and MTX in treating LPP. By comparing the effectiveness and safety profiles of these systemics, this study endeavours to provide valuable information that can guide evidence-based treatment decisions and enhance the overall understanding of LPP management.

Objective(s)

The main objective is to assess the effectiveness in routine clinical care of hydroxychloroquine (HCQ) and methotrexate (MTX) in the treatment of adults diagnosed with lichen planopilaris (LPP) by evaluating the impact on the Lichen Planopilaris Activity Index (LPPAI) after a 6-month treatment period.

Primary objective:

To investigate the difference in LPPAI between baseline and 24 weeks of treatment between the HCQ and MTX group

Secondary objectives:

2. To compare LPPAI between HCQ and MTX at 0, 12, 24, 36, and 48 weeks.

3. To compare the quality of life between HCQ and MTX at 0, 12, 24, 36, and 48 weeks.

4. To compare the side effects of HCQ and MTX.

5. To compare the proportion of patients who discontinued therapy due to sides effects in both groups.

Skindex-29

The Skindex-29 is a dermatology-specific questionnaire. It evaluates the effect of skin conditions on physical, psychological, and social aspects. It assesses the extent to which a skin condition has influenced quality of life over the past week. The 29 questions are divided into 3 domains: symptoms, emotions, and functioning. A higher score corresponds to a greater impact on quality of life.

Other disease- and treatment-related characteristics will be retrieved from the electronic patient records.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and older.
* Diagnosed with LPP.
* Willingness to provide informed consent for participation in the study.
* No contraindications or known allergies to HCQ or MTX.

Exclusion Criteria:

* Histopathological different diagnosis than LPP.
* Inability to adhere to the study protocol, including medication intake, clinic visits, and questionnaire completion.
* Patients who are ineligible for the HCQ arm (due to contraindications), are automatically included in the MTX arm.
* Contraindications HCQ:

retinopathy and/or maculopathy

myasthenia gravis

body weight less than 35 kg

Patients who are ineligible for the MTX arm (due to contraindications), are automatically included in the HCQ arm.

- Contraindications MTX:

Conception (both male and female) and lactation

Severe kidney or liver dysfunction (fibrosis, cirrhosis) or alcohol abuse

Bone marrow hypoplasia, immunodeficiency

Anemia, leukopenia, or thrombocytopenia

Poor nutritional status (low albumin)

Hypersensitivity or allergy to MTX

Lung toxicity due to MTX or significant reduction in lung function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) patients diagnosed with LPP. All patients will be recruited at the dermatology outpatient clinics in the Erasmus University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
LPPAI | at 24 weeks
  The main study parameter is the change in Lichen PlanoPilaris Activity Index (LPPAI) measured at 6 months (0-10).

SECONDARY OUTCOMES:
LPPAI | at 0, 12, 36, 48 weeks
  The main study parameter is the change in Lichen PlanoPilaris Activity Index (LPPAI) measured (0-10).
Skindex-29 | at 0, 12, 24, 36, 48 weeks
  Quality of Life
Side effects | at 0, 12, 24, 36, 48 weeks
  Number of side effects

CONTACTS AND LOCATIONS:
Overall Officials: DirkJan Hijnen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Undecided